CLINICAL TRIAL: NCT01437098
Title: Clinical Evaluation of MDT-2111 in Subjects With Symptomatic Severe Aortic Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT-2111
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Aortic Valve Stenosis
Keywords: Valvular Heart Disease; Severe Aortic Stenosis; Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MDT-2111 CoreValve TAVI (Experimental): Transcatheter Aortic Valve Implantation (TAVI) with MDT-2111 CoreValve system. Access sites for the implant include: Iliofemoral, Subclavian and Direct Aortic.
  Interventions: Device: MDT-2111 CoreValve for TAVI

INTERVENTIONS:
Device: MDT-2111 CoreValve for TAVI — CoreValve Transcatheter Aortic Valve Implantation (TAVI) using the MDT-2111 system.

SUMMARY:
The primary objective of the present trial is to demonstrate the effectiveness and safety of the MDT-2111 in the treatment of symptomatic severe aortic stenosis in subjects deemed difficult for surgical operation.

DETAILED DESCRIPTION:
Non-randomized, prospective, multicenter, single-arm trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have co-morbidities such that one cardiologist and one cardiac surgeons agree that medical factors preclude operation, based on a conclusion that the probability of death or serious morbidity exceeds the probability of meaningful improvement.
2. Subject has senile degenerative aortic valve stenosis with:

   mean gradient > 40 mmHg or jet velocity greater than 4.0 m/s by either resting or dobutamine stress echocardiogram, or simultaneous pressure recordings at cardiac catheterization (either resting or dobutamine stress), AND an initial aortic valve area of ≤ 0.8 cm² (or aortic valve area index ≤ 0.5 cm²/m²) by resting echocardiogram.
3. Subject is symptomatic from his/her aortic valve stenosis, as demonstrated by NYHA Functional Class Class III or greater. If screening committee agrees the eligibility of a patient with class II , based on medical factors, he/she can be enrolled.
4. Subject has been informed of the nature of the trial and has signed an Informed Consent Form.
5. Subject agrees to comply with specified follow-up evaluations and to return to the same investigational site where the procedure was performed.

Exclusion Criteria:

1. Evidence of an acute myocardial infarction ≤ 30 days prior to the intended treatment.
2. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to the procedure.
3. Blood dyscrasias as defined:

   * Leukopenia (WBC count < 1,000 cells/mm³)
   * Thrombocytopenia (platelet count <50,000 cells/mm³)
   * History of bleeding diathesis or coagulopathy
   * Hypercoagulable states
4. Untreated clinically significant coronary artery disease requiring revascularization.
5. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
6. Need for emergency surgery for any reason.
7. Severe ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20% as measured by resting echocardiogram.
8. Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack(TIA).
9. End stage renal disease requiring chronic dialysis.
10. GI bleeding within the past 3 months.
11. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated:

    * Aspirin
    * Ticlopidine
    * Heparin
    * Contrast media
    * Nitinol (titanium and nickel alloy)
12. Ongoing sepsis, including active endocarditis.
13. Subject refuses a blood transfusion.
14. Life expectancy < 12 months due to associated non-cardiac co-morbid conditions.
15. Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the subject from appropriate consent.
16. Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
17. Currently participating in an investigational drug or another device trial. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
18. Symptomatic carotid or vertebral artery disease.
19. Native aortic annulus size < 20 mm or > 27 mm per the screening diagnostic imaging.
20. Pre-existing prosthetic heart valve in any position.
21. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation).
22. Mitral regurgitation (moderate to severe) or severe tricuspid regurgitation.
23. Moderate to severe mitral stenosis.
24. Hypertrophic obstructive cardiomyopathy.
25. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
26. Severe basal septal hypertrophy with an outflow gradient.
27. Ascending aorta diameter > 43 mm (in case of the aortic annulus is 23-27 mm) unless the aortic annulus is 20-23 mm in which case the ascending aorta diameter > 40 mm.
28. Congenital bicuspid or unicuspid valve verified by echocardiography.
29. For patients with native coronary artery dependent circulation:

    * Sinus of valsalva width < 29 mm unless the aortic annulus is 20-23 mm, in which case the sinus of valsalva width < 27 mm, OR
    * Height of the left or right coronary sinus of valsalva (to the tubular aorta) < 15mm.
30. Femoral or iliac artery of the first choice corresponding to any one of the followings:

    * Angle at aortic root (the angle between aortic valve annulus plane and horizontal plane/vertebra) exceeds 70°.
    * Vessel diameter of femoral or iliac artery is less than 6 mm.
    * Aorta has severe calcification, excess tortuosity or severe atherosclerosis.
    * Transarterial access not able to accommodate an 18Fr sheath.
31. Subclavian artery of the second choice corresponding to any one of the followings:

    * Angle at aortic root (the angle between aortic valve annulus plane and horizontal plane/vertebra) exceeds 70° (in the case of left subclavian artery) and 30° (in the case of right subclavian artery).
    * Vessel diameter of subclavian artery is less than 6 mm.
    * Transarterial access not able to accommodate an 18Fr sheath.
32. Direct Aortic Artery as third line choice of access. Patients are excluded from Direct Aortic access if:

    * Access site is less than 6 cm from the aortic valve basal plane
    * Access site has calcification or porcelain aorta
    * Access site and delivery trajectory contain RIMA or patent RIMA graft

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2018-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Osaka University Hospital, Suita, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Saitama Medical University, Hidaka, Saitama

REFERENCES:
- [Derived] Sawa Y, Torikai K, Kobayashi J, Niinami H, Kuratani T, Maeda K, Kanzaki H, Komiyama N, Tanaka Y, Zhang A, Saito S. Midterm Outcomes With a Self-Expandable Transcatheter Heart Valve in Japanese Patients With Symptomatic Severe Aortic Stenosis. Circ J. 2017 Jul 25;81(8):1108-1115. doi: 10.1253/circj.CJ-17-0112. Epub 2017 Mar 17. PMID 28321003
- [Derived] Sawa Y, Saito S, Kobayashi J, Niinami H, Kuratani T, Maeda K, Kanzaki H, Komiyama N, Tanaka Y, Boyle A, Zhang A, Moore BJ, de Medeiros R; MDT-2111 Japan Investigators. First clinical trial of a self-expandable transcatheter heart valve in Japan in patients with symptomatic severe aortic stenosis. Circ J. 2014;78(5):1083-90. doi: 10.1253/circj.cj-14-0162. Epub 2014 Mar 21. PMID 24662399

RESULTS

PARTICIPANT FLOW:
Groups:
- MDT-2111 TAVI: Transcatheter Aortic Valve Implantation (TAVI) with MDT-2111 system.
Period: Overall Study
Arm/Group | MDT-2111 TAVI
Started | 55
30 Days | 51
6 Months | 47
12 Months | 45
24 Months | 42
36 Months | 36
Completed | 42
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: As Treated Subjects
Arm/Group | MDT-2111 TAVI
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 17
Region of Enrollment [Number; unit: participants]
  Japan | 55
NYHA Class [Number; unit: participants] — New York Heart Association Classification (NYHA) Class I Subject with cardiac disease but without resulting limitations of physical activity. Class II Subjects with cardiac disease resulting in slight limitation of physical activity. Class III Subjects with cardiac disease resulting in marked limitation of physical activity. Class IV Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  participants
    NYHA Class II | 0
    NYHA Class III | 49
    NYHA Class IV | 6
STS Score [Mean (Standard Deviation); unit: percent] — The Society of Thoracic Surgeons (STS) risk model predicts the risk of operative mortality and morbidity after adult cardiac surgery on the basis of patient demographic and clinical variables. After information has been entered on a given case, the online STS risk calculator provides a risk percentage for each of the outcomes. The risk percentage estimates the chance of a specific outcome for a patient with the indicated risk factors. A higher score indicates a higher risk. A lower score indicates a lower risk.
  percent | 8.0 (4.2)
Logistic EuroScore [Mean (Standard Deviation); unit: percent] — The European System for Cardiac Operative Risk Evaluation (EuroSCORE) is a method of calculating predicted operative mortality for patients undergoing cardiac surgery. If a risk factor is present, a weight/number is assigned. The weights are added to give an approximate percent of predicted mortality. A higher score indicates a higher risk. A lower score indicates a lower risk..
  percent | 21.5 (9.9)
Aortic Valve Area (AVA) [Mean (Standard Deviation); unit: cm²] | 0.6 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Composite Success of Improvement in New York Heart Association (NYHA) Class and a Performance Goal for Effective Orifice Area (EOA).
Description: The primary endpoint was defined as the proportion of implanted subjects with improvement of at least 1 NYHA class from baseline to 6 months and EOA greater than 1.2 cm² at 6 months.
Time Frame: baseline and 6 months
Population: All subjects implanted with the MDT-2111 device.
Measure: Number; unit: percentage of participants
Groups:
- All Implanted Subjects: The Implanted population consisted of all As Treated Subjects who underwent an index procedure and were implanted with the MDT-2111 device.
- Iliofemoral Implanted Subjects: The IF Implanted population consisted of all IF As Treated Subjects who underwent an index procedure and were implanted with the MDT-2111 device.
Arm/Group | All Implanted Subjects | Iliofemoral Implanted Subjects
Number analyzed (Participants) | 47 | 36
percentage of participants | 93.6 | 91.7
Statistical Analysis 1: Comparison: Iliofemoral Implanted Subjects; Test type: Superiority or Other; p < 0.001, Exact binomial; Proportion of IF Implanted Subjects = 91.7, 95% CI 2-sided [77.5 to 98.2]

2. Secondary Outcome: NYHA Classification Over Time
Description: NEW YORK HEART ASSOCIATION CLASSIFICATION (NYHA) Class I Subject with cardiac disease but without resulting limitations of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain.
  Class II Subjects with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III Subjects with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation, dyspnea, or anginal pain. Class IV Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 30 days
Population: NYHA denominators included deaths (n=2). Taken deaths out, you have n=51 at 30 days.
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 53
percentage of participants
  NYHA I | 58.5
  NYHA II | 30.2
  NYHA III | 5.7
  NYHA IV | 1.9
  Died prior to visit | 3.8

3. Secondary Outcome: NYHA Classification Over Time
Description: as for outcome 2
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 52
percentage of participants
  NYHA I | 59.6
  NYHA II | 30.8
  NYHA III | 0.0
  NYHA IV | 0.0
  Died prior to visit | 9.6

4. Secondary Outcome: NYHA Classification Over Time
Description: as for outcome 2
Time Frame: 12 Months
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 53
percentage of participants
  NYHA I | 60.4
  NYHA II | 24.5
  NYHA III | 0.0
  NYHA IV | 0.0
  Died prior to visit | 15.1

5. Secondary Outcome: NYHA Classification Over Time
Description: as for outcome 2
Time Frame: 24 Months
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 52
percentage of participants
  NYHA I | 59.6
  NYHA II | 21.2
  NYHA III | 0.0
  NYHA IV | 0.0
  Died prior to visit | 19.2

6. Secondary Outcome: NYHA Classification Over Time
Description: as for outcome 2
Time Frame: 36 Months
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 52
percentage of participants
  NYHA I | 57.7
  NYHA II | 9.6
  NYHA III | 0
  NYHA IV | 0
  Died prior to visit | 32.7

7. Secondary Outcome: Major Adverse Cardiovascular and Cerebrovascular Event (MACCE)
Description: MACCE is defined as a composite of:
  * all-cause death
  * myocardial infarction (MI)
  * all stroke, and
  * reintervention (defined as any cardiac surgery or percutaneous reintervention catheter procedure that repairs, otherwise alters or adjusts, or replaces a previously implanted valve)
Time Frame: 0 day to 30 days
Population: The Kaplan-Meier Method was used to calculate the number.
Measure: Number; unit: prob of freedom from event @ 30 days
Groups:
- As Treated Population: The As Treated (AT) population was defined as subjects with an attempted implant procedure, identified as subject entry to the procedure room and any of the following occurrences: anesthesia administered, vascular line placed, transesophageal echo (TEE) placed, or any monitoring line placed.
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event @ 30 days | 89.1

8. Secondary Outcome: Major Adverse Cardiovascular and Cerebrovascular Event (MACCE)
Description: as for outcome 7
Time Frame: 0 day to 6 months
Population: The Kaplan-Meier Method was used to calculate the number.
Measure: Number; unit: prob of freedom from event @ 183 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event @ 183 days | 81.6

9. Secondary Outcome: Major Adverse Cardiovascular and Cerebrovascular Event (MACCE)
Description: as for outcome 7
Time Frame: 0 day to 12 months
Population: The Kaplan-Meier Method was used to calculate the number.
Measure: Number; unit: prob of freedom from event @ 365 days
Groups:
- As Treated (AT) Population: The As Treated (AT) population was defined as subjects with an attempted implant procedure, identified as subject entry to the procedure room and any of the following occurrences: anesthesia administered, vascular line placed, transesophageal echo (TEE) placed, or any monitoring line placed.
Arm/Group | As Treated (AT) Population
Number analyzed (Participants) | 55
prob of freedom from event @ 365 days | 76.1

10. Secondary Outcome: Major Adverse Cardiovascular and Cerebrovascular Event (MACCE)
Description: as for outcome 7
Time Frame: 0 day to 24 months
Population: The Kaplan-Meier Method was used to calculate the number.
Measure: Number; unit: prob of freedom from event at 730 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event at 730 days | 68.4

11. Secondary Outcome: Major Adverse Cardiovascular and Cerebrovascular Event (MACCE)
Description: as for outcome 7
Time Frame: 0 day to 36 months
Population: The Kaplan-Meier Method was used to calculate the number.
Measure: Number; unit: prob of freedom from event at 1095 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event at 1095 days | 57.3

12. Secondary Outcome: Device Success as Defined in the Description.
Description: * successful vascular access, delivery and deployment of the device, and successful retrieval of the delivery system
  * correct position of the device in the proper anatomical location (placement in the annulus with no impedance on device function)
  * Intended performance of the prosthetic valve (aortic valve area >1.2 cm² (by echocardiography using the continuity equation) and mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/sec, without moderate or severe prosthetic valve AR)
  * Only one valve implanted in the proper anatomical location
Time Frame: after procedure or discharge
Population: The AT cohort that went through an index procedure were analyzed for Device Success. Also, all components that went into the success measures had to be non-missing. Therefore n=53.
Measure: Number; unit: percentage of participants
Groups:
- As Treated Population With Index Procedure: The As Treated (AT) population was defined as subjects with an attempted implant procedure, identified as subject entry to the procedure room and any of the following occurrences: anesthesia administered, vascular line placed, transesophageal echo (TEE) placed, or any monitoring line placed. Index procedure was defined as introduction of the MDT-2111 TAV system delivery catheter.
Arm/Group | As Treated Population With Index Procedure
Number analyzed (Participants) | 53
percentage of participants | 90.6

13. Secondary Outcome: Procedural Success, Defined as Device Success and Absence of In-hospital MACCE.
Time Frame: after procedure or discharge
Measure: Number; unit: percentage of participants
Arm/Group | As Treated Population With Index Procedure
Number analyzed (Participants) | 54
percentage of participants | 81.5

14. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Mean Gradient
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 50
mmHg | 9.5 (3.4)

15. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance- Mean Gradient
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 47
mmHg | 8.9 (2.3)

16. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Mean Gradient
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 45
mmHg | 9.4 (3.0)

17. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Mean Gradient
Time Frame: 24 months
Population: The implanted cohorts that had non-missing data at this time point were analyzed. Implanted subjects that had mean gradients available at 24 months were analyzed. Not everyone followed to 24 months had this measurement. This is true of all other echo data results, and explains if the number is different from the Number of Participants Analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 41
mmHg | 8.4 (2.6)

18. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Mean Gradient
Time Frame: 36 months
Population: The implanted cohorts that had non-missing data at this time point were analyzed. Implanted subjects that had LVEF measurement available at 36 months were analyzed. Not everyone followed to 36 months had this measurement. This is true of all other echo data results, and explains if the number is different from the Number of Participants Analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 33
mmHg | 8.9 (3.0)

19. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance- Effective Orifice Area (EOA)
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 47
cm² | 1.8 (0.4)

20. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance- Effective Orifice Area (EOA)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 47
cm² | 1.8 (0.4)

21. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance- Effective Orifice Area (EOA)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 45
cm² | 1.7 (0.4)

22. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance- Effective Orifice Area (EOA)
Time Frame: 24 months
Population: The implanted cohorts that had non-missing data at this time point were analyzed. Implanted subjects that had EOA measurement available at 24 months were analyzed. Not everyone followed to 24 months had this measurement. This is true of all other echo data results, and explains if the number is different from the Number of Participants Analyzed.
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 38
cm² | 1.8 (0.5)

23. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance- Effective Orifice Area (EOA)
Time Frame: 36 months
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 29
cm² | 1.8 (0.4)

24. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Left Ventricular Ejection Fraction (LVEF)
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 51
percent | 63.9 (6.6)

25. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Left Ventricular Ejection Fraction (LVEF)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 47
percent | 63.8 (7.7)

26. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Left Ventricular Ejection Fraction (LVEF)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 45
percent | 62.9 (7.0)

27. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Left Ventricular Ejection Fraction (LVEF)
Time Frame: 24 months
Population: The implanted cohorts that had non-missing data at this time point were analyzed. Implanted subjects that had LVEF measurement available at 24 months were analyzed. Not everyone followed to 24 months had this measurement. This is true of all other echo data results, and explains if the number is different from the Number of Participants Analyzed.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 42
percent | 64.3 (6.3)

28. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Left Ventricular Ejection Fraction (LVEF)
Time Frame: 36 months
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 35
percent | 61.1 (7.8)

29. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Total Aortic Valve Regurgitation (Transvalvular & Paravalvular) (Total AR)
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 50
percentage of participants
  None | 8.0
  Trace | 48.0
  Mild | 38.0
  Moderate | 6.0
  Severe | 0.0

30. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Total Aortic Valve Regurgitation (Transvalvular & Paravalvular) (Total AR)
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 47
percentage of participants
  None | 31.9
  Trace | 31.9
  Mild | 31.9
  Moderate | 4.3
  Severe | 0.0

31. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Total Aortic Valve Regurgitation (Transvalvular & Paravalvular) (Total AR)
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 45
percentage of participants
  None | 24.4
  Trace | 26.7
  Mild | 44.4
  Moderate | 4.4
  Severe | 0.0

32. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Total Aortic Valve Regurgitation (Transvalvular & Paravalvular) (Total AR)
Time Frame: 24 months
Population: The implanted cohorts that had non-missing data at this time point were analyzed. Implanted subjects that had Total AR available at 24 months were analyzed. Not everyone followed to 24 months had this measurement. This is true of all other echo data results, and explains if the number is different from the Number of Participants Analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 41
percentage of participants
  None | 17.1
  Trace | 41.5
  Mild | 36.6
  Moderate | 4.9
  Severe | 0.0

33. Secondary Outcome: Echocardiographic Assessment of Prosthetic Valve Performance - Total Aortic Valve Regurgitation (Transvalvular & Paravalvular) (Total AR)
Time Frame: 36 months
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 35
percentage of participants
  None | 25.7
  Trace | 31.4
  Mild | 37.1
  Moderate | 5.7
  Severe | 0.0

34. Secondary Outcome: Repeat Hospitalization
Time Frame: 0 day to 30 days
Measure: Number; unit: prob of freedom from event @ 30 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event @ 30 days | 94.3

35. Secondary Outcome: Repeat Hospitalization
Time Frame: 0 day to 6 months
Measure: Number; unit: prob of freedom from event @ 183 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event @ 183 days | 61.0

36. Secondary Outcome: Repeat Hospitalization
Time Frame: 0 day to 12 months
Measure: Number; unit: prob of freedom from event @ 365 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event @ 365 days | 50.9

37. Secondary Outcome: Repeat Hospitalization
Time Frame: 0 day to 24 months
Measure: Number; unit: prob of freedom from event @ 730 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event @ 730 days | 37.4

38. Secondary Outcome: Repeat Hospitalization
Time Frame: 0 day to 36 months
Measure: Number; unit: prob of freedom from event @ 1095 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event @ 1095 days | 35.9

39. Secondary Outcome: Valve-related Deaths
Time Frame: 0 day to 30 days
Measure: Number; unit: prob of freedom from event @ 30 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event @ 30 days | 98.2

40. Secondary Outcome: Valve-related Deaths
Time Frame: 0 day to 6 months
Measure: Number; unit: prob of freedom from event @ 183 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event @ 183 days | 98.2

41. Secondary Outcome: Valve-Related Deaths
Time Frame: 0 day to 12 months
Measure: Number; unit: prob of freedom from event @ 365 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event @ 365 days | 98.2

42. Secondary Outcome: Valve-related Deaths
Time Frame: 0 day to 24 months
Measure: Number; unit: prob of freedom from event @ 730 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event @ 730 days | 98.2

43. Secondary Outcome: Valve-related Deaths
Time Frame: 0 day to 36 months
Measure: Number; unit: prob of freedom from event @ 1095 days
Arm/Group | As Treated Population
Number analyzed (Participants) | 55
prob of freedom from event @ 1095 days | 94.5

44. Secondary Outcome: Quality of Life Assessment Using SF-36 Questionnaire - Physical Component Summary (Paired Change From Baseline) (Q of L)
Description: The SF-36 assessment was used to evaluate subject Quality of life (QoL) by assessing change in physical function and general health status. The SF-36 v2TM Scoring Program2,3 was used to convert raw scores ranging from 0 to 100 into norm-based scores, allowing direct comparison to the reference values for the Japanese population. A norm-based score of less than 50 was interpreted as below average when compared to the Japanese population whereas norm-based scores greater than 50 were interpreted as above average.
Time Frame: Baseline to 30 days
Population: The implanted cohorts that had non-missing data at this time point were analyzed. Implanted subjects that had Q of L available at this visit were analyzed. Not everyone followed to this visit had this measurement. This is true of all other echo data results, and explains if the number is different from the Number of Participants Analyzed.
Measure: Median (Inter-Quartile Range); unit: Points
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 50
Points | 5.2 [-8.1 to 18.4]

45. Secondary Outcome: Quality of Life Assessment Using SF-36 Questionnaire - Physical Component Summary (Paired Change From Baseline) (Q of L)
Description: as for outcome 44
Time Frame: Baseline to 6 months
Measure: Median (Inter-Quartile Range); unit: Points
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 47
Points | 11.2 [1.4 to 23.8]

46. Secondary Outcome: Quality of Life Assessment Using SF-36 Questionnaire - Physical Component Summary (Paired Change From Baseline) (Q of L)
Description: as for outcome 44
Time Frame: Baseline to 12 months
Measure: Median (Inter-Quartile Range); unit: Points
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 45
Points | 10.8 [-5.6 to 24.2]

47. Secondary Outcome: Quality of Life Assessment Using SF-36 Questionnaire - Physical Component Summary (Paired Change From Baseline) (Q of L)
Description: as for outcome 44
Time Frame: Baseline to 24 Months
Measure: Median (Inter-Quartile Range); unit: Points
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 41
Points | 9.3 [-5.3 to 20.1]

48. Secondary Outcome: Quality of Life Assessment Using SF-36 Questionnaire - Physical Component Summary (Paired Change From Baseline) (Q of L)
Description: as for outcome 44
Time Frame: Baseline to 36 Months
Measure: Median (Inter-Quartile Range); unit: Points
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 34
Points | 4.8 [-6.2 to 16.0]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) must be reported to the study sponsor by the investigator or study staff within 24 hours after the investigator first learns of event.
Groups:
- Iliofemoral (As Treated Subjects): The iliofemoral approach is used as the primary access site because there is a large body of clinical data in the past using this approach in patients.
- Subclavian (As Treated Subjects): The subclavian access is additionally chosen (as the secondary access site) when physicians may require an alternative to the femoral access site for patients who would benefit from the therapy but have unfavorable peripheral vasculature such as excessive atherosclerosis, calcifications, or tortuosity of common femoral arteries.
- Direct Aortic (As Treated Subjects): For patients who would benefit from the therapy but have unfavorable non-aortic vasculature of the transfemoral and subclavian/axillary access sites (i.e. excessive atherosclerosis, calcifications, or tortuosity of arteries), the direct aortic approach is currently being used in oversea(EU and US) in clinical practice with similar outcomes to transfemoral and subclavian/ axillary artery approaches.
- All Subjects (As Treated Subjects): This includes subjects from all access approaches, iliofemoral, subclavian and direct aortic.
Arm/Group | Iliofemoral (As Treated Subjects) | Subclavian (As Treated Subjects) | Direct Aortic (As Treated Subjects) | All Subjects (As Treated Subjects)
Serious Adverse Events (participants affected / at risk) | 40/44 | 4/5 | 5/6 | 49/55
Other Adverse Events (participants affected / at risk) | 44/44 | 5/5 | 6/6 | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iliofemoral (As Treated Subjects) (N=44) | Subclavian (As Treated Subjects) (N=5) | Direct Aortic (As Treated Subjects) (N=6) | All Subjects (As Treated Subjects) (N=55)
Anaemias Nec (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Aortic Valvular Disorders (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Cardiac Conduction Disorders (Cardiac disorders) | 11 (11) | 2 (2) | 0 (0) | 13 (13)
Cardiac Disorders Nec (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coronary Artery Disorders Nec (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Heart Failures Nec (Cardiac disorders) | 6 (15) | 1 (1) | 3 (6) | 10 (22)
Ischaemic Coronary Artery Disorders (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Myocardial Disorders Nec (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pericardial Disorders Nec (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Supraventricular Arrhythmias (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ventricular Arrhythmias And Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Cataract Conditions (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Gastrointestinal Ulcers And Perforation, Site Unspecified (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Non-Site Specific Gastrointestinal Haemorrhages (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 5 (5)
Asthenic Conditions (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Death And Sudden Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Device Issues Nec (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Febrile Disorders (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
General Signs And Symptoms Nec (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain And Discomfort Nec (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis And Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic Enzymes And Function Abnormalities (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic Failure And Associated Disorders (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Obstructive Bile Duct Disorders (Excl Neoplasms) (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Abdominal And Gastrointestinal Infections (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Bacterial Infections Nec (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Infections Nec (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Lower Respiratory Tract And Lung Infections (Infections and infestations) | 5 (7) | 0 (0) | 2 (5) | 7 (12)
Sepsis, Bacteraemia, Viraemia And Fungaemia Nec (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stretococcal Infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cerebral Injuries Nec (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lower Limb Fractures And Dislocations (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Non-Site Specific Injuries Nec (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-Site Specific Procedural Complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pelvic Fractures And Dislocations (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spinal Fractures And Dislocations (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Physical Examination Procedures (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diabetes Mellitus (Incl Subtypes) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
General Nutritional Disorders Nec (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle Weakness Conditions (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal And Connective Tissue Pain And Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 3 (4)
Breast And Nipple Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Hepatobiliary Neoplasms Malignancy Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Lymphomas Unspecified Nec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Central Nervous System Haemorrhages And Cerebrovascular Accidents (Nervous system disorders) | 6 (6) | 0 (0) | 2 (2) | 8 (8)
Central Nervous System Vascular Disorders Nec (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety Disorders Nec (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal Failure And Impairment (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Renal Vascular And Ischaemic Conditions (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pelvic Prolapse Conditions (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breathing Abnormalities (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower Respiratory Tract Inflammatory And Immunologic Conditions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal Disorders Nec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Parenchymal Lung Disorders Nec (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Pneumothorax And Pleural Effusions Nec (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Pulmonary Oedemas (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failures (Excl Neonatal) (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Upper Respiratory Tract Signs And Symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis Ascribed To Specific Agent (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aortic Aneurysms And Dissections (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Circulatory Collapse And Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral Embolism And Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral Vasoconstriction, Necrosis And Vascular Insufficiency (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Vascular Hypotensive Disorders (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iliofemoral (As Treated Subjects) (N=44) | Subclavian (As Treated Subjects) (N=5) | Direct Aortic (As Treated Subjects) (N=6) | All Subjects (As Treated Subjects) (N=55)
Anaemias Nec (Blood and lymphatic system disorders) | 13 (13) | 1 (2) | 2 (2) | 16 (17)
Coagulopathies (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenias (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac Conduction Disorders (Cardiac disorders) | 27 (39) | 4 (4) | 2 (3) | 33 (46)
Cardiac Signs And Symptoms Nec (Cardiac disorders) | 3 (5) | 1 (1) | 0 (0) | 4 (6)
Heart Failures Nec (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Ischaemic Coronary Artery Disorders (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mitral Valvular Disorders (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pericardial Disorders Nec (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rate And Rhythm Disorders Nec (Cardiac disorders) | 4 (4) | 0 (0) | 1 (1) | 5 (5)
Supraventricular Arrhythmias (Cardiac disorders) | 9 (11) | 0 (0) | 2 (3) | 11 (14)
Ventricular Arrhythmias And Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Ear Disorders Nec (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Inner Ear Signs And Symptoms (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Adrenal Cortical Hypofunctions (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thyroid Hypofunction Disorders (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cataract Conditions (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Excl Infective) (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (3) | 6 (7)
Gastrointestinal Atonic And Hypomotility Disorders Nec (Gastrointestinal disorders) | 7 (7) | 1 (2) | 2 (2) | 10 (11)
Gastrointestinal Inflammatory Disorders Nec (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Signs And Symptoms Nec (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea And Vomiting Symptoms (Gastrointestinal disorders) | 8 (8) | 1 (1) | 1 (2) | 10 (11)
Non-Site Specific Gastrointestinal Haemorrhages (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral Soft Tissue Disorders Nec (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tongue Disorders (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tongue Signs And Symptoms (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Administration Site Reactions Nec (General disorders) | 4 (4) | 2 (2) | 1 (2) | 7 (8)
Asthenic Conditions (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Complications Associated With Device Nec (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Febrile Disorders (General disorders) | 11 (11) | 2 (2) | 2 (2) | 15 (15)
Feelings And Sensations Nec (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Implant And Catheter Site Reactions (General disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Inflammations (General disorders) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Injection Site Reactions (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Oedema Nec (General disorders) | 8 (9) | 0 (0) | 1 (1) | 9 (10)
Pain And Discomfort Nec (General disorders) | 3 (5) | 0 (0) | 0 (0) | 3 (5)
Hepatic Enzymes And Function Abnormalities (Hepatobiliary disorders) | 2 (2) | 1 (2) | 0 (0) | 3 (4)
Bacterial Infections Nec (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infections Nec (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Infections (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Tinea Infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infections (Infections and infestations) | 5 (9) | 1 (2) | 0 (0) | 6 (11)
Urinary Tract Infections (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 4 (4)
Fractures And Dislocations Nec (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal And Hepatobiliary Procedural Complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-Site Specific Injuries Nec (Injury, poisoning and procedural complications) | 10 (10) | 1 (1) | 5 (6) | 16 (17)
Non-Site Specific Procedural Complications (Injury, poisoning and procedural complications) | 12 (16) | 0 (0) | 4 (4) | 16 (20)
Skin Injuries Nec (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0) | 4 (4)
Spinal Fractures And Dislocations (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood Counts Nec (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Coagulation And Bleeding Analyses (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Faecal Analyses Nec (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Heart Rate And Pulse Investigations (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lipoprotein And Lipid Tests Nec (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Liver Function Analyses (Investigations) | 12 (16) | 1 (1) | 2 (2) | 15 (19)
Metabolism Tests Nec (Investigations) | 5 (6) | 0 (0) | 3 (4) | 8 (10)
Mineral And Electrolyte Analyses (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Physical Examination Procedures (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Platelet Analyses (Investigations) | 10 (10) | 1 (1) | 1 (1) | 12 (12)
Protein Analyses Nec (Investigations) | 29 (31) | 3 (3) | 2 (2) | 34 (36)
Red Blood Cell Analyses (Investigations) | 6 (6) | 0 (0) | 0 (0) | 6 (6)
Renal Function Analyses (Investigations) | 3 (3) | 1 (1) | 1 (1) | 5 (5)
Skeletal And Cardiac Muscle Analyses (Investigations) | 12 (15) | 3 (3) | 6 (7) | 21 (25)
Tissue Enzyme Analyses Nec (Investigations) | 7 (10) | 0 (0) | 3 (3) | 10 (13)
Triglyceride Analyses (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Urinary Tract Function Analyses Nec (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Vascular Tests Nec (Incl Blood Pressure) (Investigations) | 14 (19) | 2 (2) | 3 (4) | 19 (25)
White Blood Cell Analyses (Investigations) | 12 (12) | 3 (3) | 0 (0) | 15 (15)
Appetite Disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Diabetes Mellitus (Incl Subtypes) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Disorders Of Purine Metabolism (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
General Nutritional Disorders Nec (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemic Conditions Nec (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Potassium Imbalance (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 1 (1) | 6 (6)
Protein Metabolism Disorders Nec (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 2 (2) | 7 (7)
Total Fluid Volume Decreased (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Connective Tissue Disorders (Excl Le) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint Related Disorders Nec (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal And Connective Tissue Pain And Discomfort (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 1 (1) | 7 (7)
Musculoskeletal And Connective Tissue Signs And Symptoms Nec (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Soft Tissue Disorders Nec (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Tendon Disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Central Nervous System Haemorrhages And Cerebrovascular Accidents (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cortical Dysfunction Nec (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headaches Nec (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Neurological Signs And Symptoms Nec (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paralysis And Paresis (Excl Cranial Nerve) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sensory Abnormalities Nec (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vagus Nerve Disorders (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety Disorders Nec (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety Symptoms (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depressive Disorders (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Disturbances In Initiating And Maintaining Sleep (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Increased Physical Activity Levels (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal Failure And Impairment (Renal and urinary disorders) | 5 (5) | 1 (1) | 2 (2) | 8 (8)
Urinary Abnormalities (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Breast Disorders Nec (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breast Signs And Symptoms (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Vulvovaginal Disorders Nec (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breathing Abnormalities (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 4 (5)
Coughing And Associated Symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Nasal Disorders Nec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Pneumothorax And Pleural Effusions Nec (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4)
Pulmonary Oedemas (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Respiratory Failures (Excl Neonatal) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Signs And Symptoms (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Dermal And Epidermal Conditions Nec (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis And Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 5 (5)
Dermatitis Ascribed To Specific Agent (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Erythemas (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Exfoliative Conditions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratoses (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ichthyoses (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus Nec (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Purpura And Related Conditions (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin And Subcutaneous Tissue Ulcerations (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Skin Haemorrhages (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Skin Injuries And Mechanical Dermatoses (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 2 (4)
Aortic Aneurysms And Dissections (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood Pressure Disorders Nec (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Haemorrhages Nec (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-Site Specific Necrosis And Vascular Insufficiency Nec (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral Aneurysms And Dissections (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Peripheral Vasoconstriction, Necrosis And Vascular Insufficiency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vascular Hypotensive Disorders (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Vascular Malformations And Acquired Anomalies (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is not required per Japan GCP. There is an agreement with the site, but not the individual investigator at the site.